CLINICAL TRIAL: NCT03168828
Title: A Prospective, Multi-center, Open-label Study of Trospium Delivered Intravesically by TAR-302-5018 to Spinal Cord Injury Subjects With Neurogenic Detrusor Overactivity (NDO)
Brief Title: Safety and Tolerability of TAR-302-5018 in Subjects With Neurogenic Detrusor Overactivity Resulting From Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taris Biomedical LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAR-302-101
Record Dates: First submitted 2017-04-06; First posted 2017-05-30 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Neurogenic Detrusor Overactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAR-302-5018 (Experimental): Trospium-Releasing Intravesical System (TAR-302-5018) is placed into the bladder through an inserter on Study Day 0 and is removed on Study Day 42. TAR-302-5018 releases trospium gradually during the 42 day indwelling time.
  Interventions: Drug: Trospium-Releasing Intravesical System (TAR-302-5018)

INTERVENTIONS:
Drug: Trospium-Releasing Intravesical System (TAR-302-5018) — TAR-302-5018 is a passive, nonresorbable trospium-releasing intravesical system whose primary mode of action is the controlled release of trospium into the bladder over a 42-day period.

SUMMARY:
The purpose of this study is to determine if TAR-302-5018, an investigational drug-delivery system, is safe and tolerable in patients with neurogenic detrusor overactivity (NDO) resulting from spinal cord injury (SCI).

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of traumatic or nontraumatic suprasacral SCI for longer than 6 months and a documented history of NDO.
2. Age ≥ 18 years.
3. Demonstrated competence in and currently uses intermittent catheterization (IC) to empty the bladder (minimum of 4 IC events/day).

   * No indwelling catheter permitted
   * Caregiver may perform IC
   * Subject must be willing to maintain an established IC frequency throughout the study
4. History of non-stress-based urinary incontinence.

Exclusion Criteria

1. Participation in another drug or device study within 60 days prior to the screening visit.
2. Previous urologic surgery that either decreases outlet resistance (transurethral prostatectomy, urethral stent, sphincterotomy) or changes native bladder anatomy (bladder augmentation).
3. Presence of significant renal dysfunction at screening (Glomerular Filtration Rate < 30 mL/min).
4. Presence of significant polyuria of any cause at screening (urine output > 4,000 mL/day).
5. History of pelvic radiation.
6. History of either bladder cancer or bladder pathology that the investigator deems unfit for study inclusion.
7. Active malignancies within 12 months with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome.
8. Symptomatic autonomic dysreflexia requiring ongoing treatment.
9. In the opinion of the investigator, the subject has a history of significant stress urinary incontinence.
10. Subjects with active bladder stones or history of bladder stones < 6 months prior to study entry.
11. History of recurrent symptomatic UTIs (> 6 per 1 year).
12. Subjects with either untreated urinary retention or gastric retention or uncontrolled narrow-angle glaucoma.
13. Subjects with known hypersensitivity to trospium or chemically-related drugs.
14. Subjects with known hypersensitivity to nitinol or silicone.
15. Subjects actively taking oral trospium. If previously used and discontinued, these medications must have been stopped for >2 weeks.
16. The addition of a new or a change in dose to a current medication for the treatment of OAB (i.e. anticholinergics, beta-3 adrenergic agonists, antispasmodics, antidepressants, or hormones) within 30 days prior to signing the Informed Consent Form (ICF). A current dose must continue through the final study visit. If previously used and discontinued, these medications must have been stopped for > 2 weeks prior to Day 0.
17. Intravesical onabotulinum toxin use within the last 9 months prior to the screening visit.
18. Intravesical anticholinergic medications within the last 30 days prior to the screening visit.
19. History of non-medication based therapy (i.e. Interstim therapy) for the treatment of OAB. History of non-invasive neuromodulation (i.e. Percutaneous Tibial Nerve Stimulation (PTNS)) is allowed if discontinued at least 8 weeks prior to Study Day 0.
20. Female subject who is pregnant (as verified by urine test at time of screening) or lactating or of childbearing potential and not using acceptable methods of contraception.
21. Subject has a medical condition that may cause noncompliance with the study protocol.
22. Subject refuses to provide written informed consent.
23. Subject will be unable or unwilling to complete the questionnaires, diaries, or attend all protocol mandated study visits.
24. Presence of any bladder or urethral anatomic feature that in the opinion of the investigator may prevent the safe placement, indwelling use or removal of TAR-302-5018.
25. History or presence of any significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, gynecological, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder that, in the opinion of the investigator, contraindicates participation.
26. History of any of the following within 3 months prior to Screening Visit:

    1. Major illness/major surgery (requiring hospitalization), including pelvic, lower back surgery or procedure unrelated to bladder cancer; most outpatient procedures are not exclusionary
    2. Renal or ureteral stone disease or instrumentation
    3. Childbirth
27. Difficulty providing blood samples.
28. Other unspecified reasons that, in the opinion of the investigator or TARIS, make the subject unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Safety of TAR-302-5018: Safety will be assessed throughout the study based on reported AEs | Safety will be assessed from the signing of the informed consent form through Study Day 49 (+ 7 days) for a total of up to 77 days.
  Safety will be assessed throughout the study based on reported AEs, investigational product events (IPEs), physical examinations (PEs), vital signs, clinical laboratory tests, scheduled cystoscopic examinations, bladder ultrasounds, bladder post-void residual volume (PVR), and the use of concomitant medications.

SECONDARY OUTCOMES:
Tolerability of TAR-302-5018 | Tolerability will be assessed during the 42-day indwelling period unless removed due to lack of tolerability in advance of the Day 42 scheduled removal.
  Tolerability will be determined by the proportion of subjects who require TAR-302-5018 removal prior to the planned removal on Day 42 due to meeting any of the Subject Stopping Safety Criteria or other drug or device constituent related adverse event.
Peak Plasma Concentration (Cmax) | Seven time-points across 49 days (Day 0 through Day 49).
  Plasma will be evaluated for trospium levels on Study Days 0, 3, 7, 14, 28, 42, and 49.
Peak Urine Concentration (Cmax) | Seven time-points across 49 days (Day 0 through Day 49).
  Urine will be evaluated for trospium levels on Study Days 0, 3, 7, 14, 28, 42, and 49.
Preliminary Urodynamic Efficacy: Vesical Filling Phase - Instillation Volume | Day 0, Day 14 (+/- 1 day), Day 42
  Instillation volume at first sensation (mL)
Preliminary Urodynamic Efficacy: Vesical Filling Phase - Vesical Pressure | Day 0, Day 14 (+/- 1 day), Day 42
  Vesical pressure at first sensation (cmH2O)
Preliminary Urodynamic Efficacy: Vesical Filling Phase - Instillation Volume | Day 0, Day 14 (+/- 1 day), Day 42
  Instillation volume at first desire to urinate (mL)
Preliminary Urodynamic Efficacy: Vesical Filling Phase - Vesical Pressure | Day 0, Day 14 (+/- 1 day), Day 42
  Vesical pressure at first desire to urinate (cmH2O)
Preliminary Urodynamic Efficacy: Vesical Filling Phase - Instillation Volume | Day 0, Day 14 (+/- 1 day), Day 42
  Instillation volume at maximal desire to urinate (mL)
Preliminary Urodynamic Efficacy: Vesical Filling Phase - Vesical Pressure | Day 0, Day 14 (+/- 1 day), Day 42
  Vesical pressure at maximal desire to urinate (cmH2O)
Preliminary Urodynamic Efficacy: Vesical Filling Phase - Instillation Volume | Day 0, Day 14 (+/- 1 day), Day 42
  Instillation volume at maximum capacity (mL)
Preliminary Urodynamic Efficacy: Vesical Filling Phase - Detrusor Pressure | Day 0, Day 14 (+/- 1 day), Day 42
  Detrusor pressure at maximum capacity (cmH2O)
Preliminary Urodynamic Efficacy: Vesical Filling Phase - Bladder Compliance | Day 0, Day 14 (+/- 1 day), Day 42
  Bladder compliance (mL/cmH2O)
Preliminary Urodynamic Efficacy: Involuntary Bladder Contractions - Instillation Volume | Day 0, Day 14 (+/- 1 day), Day 42
  Instillation Volume (mL)
Preliminary Urodynamic Efficacy: Involuntary Bladder Contractions - Vesical Pressure | Day 0, Day 14 (+/- 1 day), Day 42
  Vesical pressure (cmH2O)
Preliminary Urodynamic Efficacy: Involuntary Bladder Contractions - Detrusor Pressure | Day 0, Day 14 (+/- 1 day), Day 42
  Detrusor pressure (cmH2O)
Preliminary Urodynamic Efficacy: Vesical Voiding Phase - Peak Flow | Day 0, Day 14 (+/- 1 day), Day 42
  Peak flow (mL/s)
Preliminary Urodynamic Efficacy: Vesical Voiding Phase - Mean Flow | Day 0, Day 14 (+/- 1 day), Day 42
  Mean flow (mL/s)
Preliminary Urodynamic Efficacy: Vesical Voiding Phase - Detrusor Pressure | Day 0, Day 14 (+/- 1 day), Day 42
  Detrusor pressure at the peak flow (cmH2O)
Preliminary Urodynamic Efficacy: Vesical Voiding Phase - Total Voided Volume | Day 0, Day 14 (+/- 1 day), Day 42
  Total voided volume (mL)
Preliminary Urodynamic Efficacy: Vesical Voiding Phase - Post Void Residual Volume | Day 0, Day 14 (+/- 1 day), Day 42
  Post void residual volume (mL)

OTHER OUTCOMES:
The Change in Quality of Life as assessed by Qualiveen Surveys | Three time-points across 42 days (Study Day 0 to Study Day 42).
  Evidence of improvement in QoL assessed at Study Days 14 (± 1 day) and 42 and compared to Study Day 0 (baseline) as assessed by the following instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kennelly, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - Michigan Institute of Urology, Troy, Michigan
  - Carolinas HealthCare System, Charlotte, North Carolina
  - Urology of Virginia, Virginia Beach, Virginia
  - Virginia Mason, Seattle, Washington